CLINICAL TRIAL: NCT06142708
Title: The Effect of Dual Trigger (GnRH Agonist + hCG) for Final Maturation in Oocyte Donors With History of a Previous Cycle With Suboptimal Response to GnRH Agonist Only Trigger
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Embryolab Fertility Clinic (Other)
Collaborators: ART Fertility Clinics LLC (Other)
Responsible Party: Principal Investigator, Nikolaos Christoforidis, Consultant Obstetrician Gynaecologist - Clinical Director, Embryolab Fertility Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 012023
Record Dates: First submitted 2023-11-09; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Ovarian Stimulation; Human Chorionic Gonadotropin; Oocyte Donors
Keywords: GnRH agonist; Dual trigger; Oocyte Donors
MeSH Terms: interventions — Chorionic Gonadotropin; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual trigger (GnRH-agonist plus hCG) (Experimental): Participants in this arm will be administered a GnRH-agonist trigger plus hCG (dual trigger) for final maturation
  Interventions: Drug: Dual trigger (human chorionic gonadotropin plus GnRH-agonist)
- Gn-RH-agonist only trigger (Active Comparator): Participants in this arm will be administered a GnRH-agonist trigger only for final maturation
  Interventions: Drug: GnRH-agonist only trigger

INTERVENTIONS:
Drug: Dual trigger (human chorionic gonadotropin plus GnRH-agonist) — Human chorionic gonadotropin will be added to GnRH-agonist as a dual trigger in participants previously having had a suboptimal response to GnRH-agonist trigger only
  Arms: Dual trigger (GnRH-agonist plus hCG)
Drug: GnRH-agonist only trigger — GnRH-agonist only will be used for final maturation
  Arms: Gn-RH-agonist only trigger

SUMMARY:
The goal of this clinical trial is to compare GnRH-agonist trigger with dual GnRH-agonist and HCG trigger in oocyte donors.

The main questions it aims to answer are:

* Maturation rate (Metaphase II/ Total number of COCs collected)
* Fertilization rate
* Embryo quality day 3
* Fragmentation rate embryo day 3
* Blastulation rate (Day5/6/7)
* Quality of blastocyst (Gardner criteria) Participants will undergo controlled ovarian stimulation with a GnRH antagonist protocol Researchers will compare the effects of final maturation with GnRH-agonist trigger to a dual trigger (hCG and GnRH-a)

DETAILED DESCRIPTION:
Final oocyte maturation is a critical step in the process of the Assisted Reproductive Technology (ART) treatment and has a certain impact on oocyte yield and oocyte competency. There are three different types of trigger: hCG, GnRH-agonist or dual trigger (hCG and GnRH-agonist combined), and the choice depends on the ovarian stimulation protocol, the ovarian response and on the clinical standard of the IVF clinic. As oocyte donors are at high risk for OHSS, a GnRH-agonist trigger (GnRH-a) is the most commonly used modality for triggering final maturation. However, a certain number of oocyte donors may have a suboptimal response to GnRH-a trigger only, with a yield of oocytes less than the 10th percentile, with a clear negative impact on oocyte efficiency and competency. This study aims to evaluate whether oocyte competence can be improved in oocyte donors with a previously suboptimal response to GnRH-a, by using a dual trigger in a subsequent ovarian stimulation cycle, in which hCG is added to the GnRH-agonist for final maturation

ELIGIBILITY:
Inclusion Criteria:

* BMI: 18 - 25
* AMH: 1-3ng/ml
* AFC: 15
* Peak E2 in previous ovarian stimulation cycle: < 4000 pg/ml
* Ovarian response in first stimulation cycle: < 20 follicles over 10mm in total, at time of triggering
* Peak E2 in study cycle: < 4000 pg/ml
* Suboptimal response to trigger medication at first stimulation cycle
* Male age < 50 years old with normospermia

Exclusion Criteria:

* Oocyte donors which are at risk for development of ovarian hyperstimulation syndrome (OHSS)

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Oocyte donors in IVF treatment
Enrollment: 80 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Oocyte maturation rate | 18 months prospective trial
  Number of metaphase II oocytes per total number of oocytes retrieved in oocyte pick-up day
Fertilization rate | 18 months prospective trial
  number of 2PN embryos per total number of MII oocytes fertilised
Blastulation rate | 18 months prospective trial
  Number of blastocysts up to day 6 per number of fertilised 2PN embryos

SECONDARY OUTCOMES:
Number of recipients per donor cycle | 18 months prospective trial
  The number of recipients matched per donor
Ongoing Pregnancy Rate | 28 months prospective trial
  number of pregnancies with positive fetal heart per number of embryotransfers performed
Live Birth Rate | 28 months prospective trial
  number of live births per number of embryotransfers performed

CONTACTS AND LOCATIONS:
Locations (1):
- Embryolab Fertility Clinic, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Yes
At the trial completion IPD are to be shared with researchers from ART Fertility Clinics for statistical analysis
Supporting Information: Study Protocol, SAP
Time Frame: at the end of study as already submitted